CLINICAL TRIAL: NCT06564831
Title: A Randomized Controlled Multicenter Clinical Trial, Evaluating the Efficacy of a Single Layer Placental-based Allograft and Standard of Care Versus Standard of Care Alone in the Management of Nonhealing Diabetic Foot Ulcers
Brief Title: Evaluating the Efficacy of a Single Layer Placental-based Allograft and Standard of Care Versus Standard of Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Biologics, LLC (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMPX
Record Dates: First submitted 2024-08-15; First posted 2024-08-21 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot; Foot Ulcer; Ulcer Foot; DFU
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer

STUDY DESIGN:
Intervention Model Description: The study will evaluate the efficacy of a single layer amniotic membrane (SLAM) and standard of care (SOC) versus SOC alone in the closure of nonhealing diabetic foot ulcers (DFUs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Other: Standard of Care Standard of care will be cleaning, debridement, ulcer moisture balance, and offloading.
  Interventions: Other: SOC
- SLAM + SOC (Experimental): Single layer amniotic membrane (SLAM) + SOC
  Interventions: Other: SLAM + SOC

INTERVENTIONS:
Other: SLAM + SOC — Weekly Treatment visits for 12 weeks begin at day 0. SLAM applications with SOC until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: SLAM + SOC
Other: SOC — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Standard of Care

SUMMARY:
A Randomized Controlled Multicenter Clinical Trial, Evaluating the Efficacy of a Single Layer Placental-based Allograft and Standard of Care versus Standard of Care alone in the management of Nonhealing Diabetic Foot Ulcers

DETAILED DESCRIPTION:
XCAMP is a multi-center randomized controlled clinical trial. The study will evaluate the efficacy of a single layer amniotic membrane (SLAM) and standard of care (SOC) versus SOC alone in the closure of nonhealing diabetic foot ulcers (DFUs). XWRAP® is an allograft membrane derived from human amniotic tissue. Designed to act as a protective barrier, it is effective for DFUs, venous leg ulcers (VLUs), and pressure ulcers [13]. The processing of XWRAP® is designed to preserve the structural integrity of the amniotic epithelial membrane [13]. The product is screened and tested in a Clinical Laboratory Improvement Amendment (CLIA) certified lab that meets or exceeds AATB criteria [13].

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age or older,
2. Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
3. At randomization subjects must have a target ulcer with a minimum surface area of 0.7 cm2 and a maximum surface area of 20.0 cm2 measured post debridement.
4. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
6. The target ulcer must be Wager 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle, provided it is below the medial aspect of the malleolus. The ulcer may not include exposed tendon or bone.
7. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. ABI ≥ 0.7 and ≤ 1.3;
   2. TBI ≥ 0.6;
   3. TCOM ≥ 40 mmHg;
   4. PVR: biphasic.
8. If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. The subject must consent to using the prescribed off-loading method for the duration of the study.
10. The subject must agree to attend the weekly study visits required by the protocol.
11. The subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

1. A subject known to have a life expectancy of < 6 months is excluded.
2. The subject is excluded if the target ulcer is not secondary to diabetes.
3. If the target ulcer is infected or if there is cellulitis in the surrounding skin, the subject is excluded.
4. If there is evidence of osteomyelitis complicating the target ulcer, the subject is excluded.
5. A potential subject cannot have an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
6. A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy is excluded.
7. The topical application of steroids to the ulcer surface within one month of initial screening is not permitted.
8. A subject with a previous partial amputation on the affected foot is excluded if the resulting deformity impedes proper offloading of the target ulcer.
9. The potential subject has a glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
10. The subject is excluded if the surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). Photographic planimetry is not required for measurements taken during the historical run-in period (e.g. calculating surface area using length x width is acceptable).
11. The subject is excluded if the surface area measurement of the Target ulcer decreases by 20% or more during the 2-week screening phase: the 2 weeks from the initial screening visit (S1) to the TV-1/randomization visit during which time the subject received SOC.
12. A subject with an acute Charcot foot, or an inactive Charcot foot, that impedes proper offloading of the target ulcer is excluded.
13. Women who are pregnant or considering becoming pregnant within the next 6 months are excluded.
14. A potential subject with end stage renal disease requiring dialysis is excluded.
15. A subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments is excluded.
16. A Subject treated with hyperbaric oxygen therapy or a Cellular and/or Tissue Product (CTP) in the 30 days prior to the initial screening visit is excluded.
17. The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The percentage of target ulcers achieving complete wound closure in 12 weeks. | 1-12 Weeks
  The percentage of target ulcers achieving complete wound closure in 12 weeks.

SECONDARY OUTCOMES:
The time to heal for target ulcers. | 1-12 weeks
  Time to closure will be determined for each treatment group and compared to SOC.
Wound Area Reduction | 1-12 weeks
  Percentage wound area reduction from TV-1 to TV-13 measured weekly with digital photographic planimetry, using MolecuLight Imaging Device, and physical examination.
Adverse Events | 1-14 Weeks
  Incidence of adverse events will be evaluated weekly from TV-1 to the healing confirmation visit (HCV).
Change in pain in the target ulcer | 1-12 weeks
  Change in pain in the target ulcer assessed using the PEG (pain, enjoyment in life, and general pain) scale. [Time Frame: TV-1, 3 weeks, 6 weeks, 9 weeks, and 12 weeks or Final Visit].
Change in quality of life | 1-12 weeks
  Change in quality-of-life using the wQOL(Wound Quality of Life) questionnaire [Time Frame: TV-1, 3 weeks, 6 weeks, 9 weeks, and 12 weeks or Final Visit].

OTHER OUTCOMES:
Percentage of target ulcers achieving complete wound closure | 1-12 weeks
  Percentage of target ulcers achieving complete wound closure in 12 weeks for subjects 65 years of age or older.
Changes in chronic inhibitory bacterial load | 1-14 weeks
  Changes in chronic inhibitory bacterial load (CIBL) measured using fluorescence imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Detroit Foot and Ankle, Clinton Township, Michigan, United States

IPD SHARING:
Plan to Share IPD: No